CLINICAL TRIAL: NCT01908166
Title: US Elastography for Characterizing Focal Lesions in the Liver and Kidney
Brief Title: Ultrasound Elastography in Diagnosing Patients With Kidney or Liver Solid Focal Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Juergen Willmann, Professor of Radiology, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: VAR0099; NCI-2013-01353 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P30CA124435 (NIH)
Record Dates: First submitted 2013-07-23; First posted 2013-07-25 (Estimated); Last update posted 2017-06-08 (Actual); Status verified 2017-06

CONDITIONS: Adult Primary Liver Cancer; Kidney Tumor
MeSH Terms: conditions — Carcinoma, Hepatocellular; Carcinoma, Renal Cell

ARMS (1):
- Diagnostic (ultrasound elastography) (Experimental): Patients undergo ultrasound elastography.
  Interventions: Procedure: ultrasound elasticity imaging

INTERVENTIONS:
Procedure: ultrasound elasticity imaging — Undergo ultrasound elastography

SUMMARY:
This clinical trial studies ultrasound elastography in diagnosing patients with kidney or liver solid focal lesions. New diagnostic procedures, such as ultrasound elastography, may be a less invasive way to check for kidney or liver solid focal lesions.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the utility of ultrasound elastography in correlation with kidney or liver biopsy or magnetic resonance imaging (MRI) or computed tomography (CT) results.

OUTLINE:

Patients undergo ultrasound elastography.

ELIGIBILITY:
Inclusion Criteria:

* There are no restrictions on life expectancy
* Eastern Cooperative Oncology Group (ECOG) or Karnofsky performance status will not be employed
* Patients of any ethnic background
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients should not be taking other investigational agents
* No requirements due to co-morbid disease or intercurrent illness, as needed
* No restrictions on allergic reactions as no imaging agent will be used
* Concomitant medications for treatment of the target lesion
* Pregnant or nursing patients will be excluded from the study

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2014-01; Primary Completion 2016-11-01 (Actual); Study Completion 2016-11-01 (Actual)

PRIMARY OUTCOMES:
Strain ratio for all lesions measured by comparing the lesion to the adjacent normal tissue | Up to 36 months
  Suspicious liver and kidney lesions will be analyzed separately on a per-lesion basis. Within each population, the strain ratio of cases and controls will be compared using the Wilcoxon rank sum test, and the analysis will be illustrated using the non-parametric receiver operating characteristic (ROC).

CONTACTS AND LOCATIONS:
Overall Officials: Juergen Willmann, Principal Investigator — Stanford University Hospitals and Clinics
Locations (1):
- Stanford University, School of Medicine, Stanford, California, United States